CLINICAL TRIAL: NCT03431584
Title: Effects on the Pain of an Infiltration by Acid Hyaluronic Association and Corticoids Versus Only Corticoids in the Rhizarthrosis.
Acronym: RHIZ'ART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHD 046-17
Record Dates: First submitted 2018-02-06; First posted 2018-02-13 (Actual); Results first posted 2025-09-29 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Rhizarthrosis
MeSH Terms: interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infiltration of corticosteroids (Active Comparator)
  Interventions: Drug: infiltration of corticosteroids
- Infiltration of corticosteroids and hyaluronic acid (Experimental)
  Interventions: Drug: infiltration of corticosteroids and hyaluronic acid

INTERVENTIONS:
Drug: infiltration of corticosteroids — infiltration of corticosteroids
  Arms: Infiltration of corticosteroids
Drug: infiltration of corticosteroids and hyaluronic acid — infiltration of corticosteroids and hyaluronic acid
  Arms: Infiltration of corticosteroids and hyaluronic acid

SUMMARY:
The rhizarthrosis, or the degenerative osteoarthritis of the trapezo-metacarpal joint, is a frequent degenerative osteoarthritis.

The treatment associates not pharmacological measures, such as resting relative of the joint, the orthosis of rest, glazing and pharmacological measures such analgesic, anti-inflammatory not steroidal per bones or premises, even infiltrations cortisone or by hyaluronic acid.

No study has, for the moment, tested the interest of the combination of cortisone and hyaluronic acid in rhizarthrosis. In view of the current publications, we propose to carry out a study on two arms, with corticosteroids in reference arm; the experimental arm is the combination of hyaluronic acid and cortisone.

ELIGIBILITY:
Inclusion Criteria:

* Adults, ≥ 40 years
* Pain located at the root of the thumb (near the wrist) and awakened by direct pressure and movement
* Pain resistant to well-conducted medical treatment, with analgesics, NSAIDs, icing with pain (analog visual scale) ≥ 4 for more than 3 months
* Radiological findings (kapandji face + profile incidence) typical of rhizarthrosis, stage II or III of Eaton and Litter, with at least 2 of the following 5 radiological elements observed on the trapeziometacarpal joint:

  * marginal osteophyte
  * pinching of the joint space
  * sclerosis of the subchondral space
  * subchondral kyst
  * absence of osteopenia
* Patient with the ability to understand the protocol and signed informed consent
* Patient receiving social security

Exclusion Criteria:

* Known allergy to any of the products (corticosteroids or hyaluronic acid) including its excipients (methyl parahydroxybenzoate, propyl parahydroxybenzoate, benzyl alcohol)
* Change of analgesic treatment within 4 weeks before inclusion.
* Patients with symptomatic bilateral rhizarthrosis
* Scaphoid-trapezial arthrosis
* Local or general infection
* Severe coagulation disorders, ongoing anticoagulant therapy
* severe and / or uncontrolled hypertension
* Earlier local surgery
* Associated inflammatory rheumatism
* Tendinopathy of De Quervain, thumb to jump associated
* Infiltrations earlier than 6 months
* Diabetes imbalanced
* Live vaccines
* Severe water and / or sodium retention (hypernatremia), particularly in cases of heart failure, decompensated liver failure (edema and ascites failure)
* Pregnant or lactating women
* Immunocompromised or hemodialysis patients
* Patients under guardianship, trusteeship, or deprived of liberty
* Patients participating in another clinical research protocol involving a drug or medical device
* Patients unable to follow the protocol, according to the judgment of the investigator

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-12-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CH Cholet, Cholet
  - CHD Vendée, La Roche-sur-Yon
  - CH Le Mans, Le Mans
  - CHU Nantes, Nantes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cormier G, Le Goff B, Denis A, Varin S, Auzanneau L, Dimet J, Le Thuaut A. Corticosteroids injections versus corticosteroids with hyaluronic acid injections in rhizarthrosis: the randomised multicentre RHIZ'ART trial study protocol. BMJ Open. 2019 Jan 9;9(1):e022553. doi: 10.1136/bmjopen-2018-022553. PMID 30782680
- [Result] Cormier G, Denis A, Leske C, Varin S, Dimet J, Planche L, Le Goff B. Improvement of rhizarthrosis pain management with the infiltration of hyaluronic acid and corticosteroids versus corticosteroids alone. Joint Bone Spine. 2025 Jul;92(4):105849. doi: 10.1016/j.jbspin.2025.105849. Epub 2025 Jan 30. PMID 39892589

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 150 patients were randomised, 1 patient was excluded from follow-up after infiltration before the first visit at M1 and was not analysed.
Period: Overall Study
Arm/Group | Infiltration of corticosteroids and hyaluronic acid | Infiltration of corticosteroids
Started | 74 | 76
Completed | 65 | 69
Not Completed | 9 | 7

BASELINE CHARACTERISTICS:
Population: One patient was lost to follow-up after infiltration and was not included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Infiltration of Corticosteroids | Infiltration of Corticosteroids and Hyaluronic Acid | Total
Number analyzed (Participants) | 76 | 73 | 149
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62 (9) | 62 (9) | 62 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 61 | 123
  Male | 14 | 12 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Analogical Visual Scale of Pain (VAS)
Description: Analogical visual scale of pain (VAS) To 0 cm (no pain) form 10 cm (worst pain imaginable)
Time Frame: 3 month post infiltration
Measure: Least Squares Mean (95% Confidence Interval); unit: centimeter
Arm/Group | Infiltration of corticosteroids | Infiltration of corticosteroids and hyaluronic acid
Number analyzed (Participants) | 73 | 73
centimeter | -1.66 [-2.29 to -1.03] | -2.65 [-3.29 to -2.01]

ADVERSE EVENTS:
Time Frame: Through study completion, , an average of 1 year
Arm/Group | Infiltration of corticosteroids | Infiltration of corticosteroids and hyaluronic acid
All-Cause Mortality (participants affected / at risk) | 1/76 | 0/73
Serious Adverse Events (participants affected / at risk) | 16/76 | 11/73
Other Adverse Events (participants affected / at risk) | 13/76 | 10/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infiltration of corticosteroids (N=76) | Infiltration of corticosteroids and hyaluronic acid (N=73)
LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OVARIAN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PYOGENIC GRANULOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
JOINT ARTHROPLASTY (Surgical and medical procedures) | 1 (1) | 0 (0)
TRAPEZIECTOMY (Surgical and medical procedures) | 2 (2) | 0 (0)
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 1 (1) | 2 (2)
PYREXIA (General disorders) | 1 (1) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
ALCOHOL ABUSE (Psychiatric disorders) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
TENOSYNOVITIS STENOSANS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infiltration of corticosteroids (N=76) | Infiltration of corticosteroids and hyaluronic acid (N=73)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (13) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/84/NCT03431584/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/84/NCT03431584/ICF_001.pdf